CLINICAL TRIAL: NCT02476981
Title: Comparison of Remifentanil and Dexmedetomidine for Monitored Anaesthesia Care
Brief Title: Comparison of Remifentanil and Dexmedetomidine for Monitored Anaesthesia Care During Vertebroplasty and Kyphoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-I039
Record Dates: First submitted 2015-06-16; First posted 2015-06-22 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Fractures, Compression
MeSH Terms: conditions — Fractures, Compression | interventions — Remifentanil; Dexmedetomidine; Midazolam; Propofol; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Remifentanil (Experimental): Remifentanil is commonly used in monitored anesthesia care because of its rapid onset and short duration of action.
  Interventions: Drug: Remifentanil
- Dexmedetomidine (Experimental): Dexmedetomidine is a highly selective α 2 adrenergic agonist and has both sedative and analgesic properties, and rarely causes respiratory depression.
  Interventions: Drug: Dexmedetomidine
- midazolam (Other): Midazolam is commonly used before induction for its anxiolytic effect.
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine; Drug: midazolam
- propofol (Other): Propofol is the most commonly used in sedative analgesia for its rapid onset and recovery time.
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine; Drug: propofol
- ephedrine (Other): Adrenergic agonist to treat hypotension
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine; Drug: ephedrine

INTERVENTIONS:
Drug: Remifentanil — Patients given remifentanil received continuous infusion of the drug at 1-5 µg/kg/h
  Other Names: Ultiva
  Arms: Remifentanil; ephedrine; midazolam; propofol
Drug: Dexmedetomidine — Patients receiving dexmedetomidine were given that drug at 0.3-0.4 µg/kg over 10 min, followed by continuous infusion of 0.2 1 µg/kg/h
  Other Names: Precedex
  Arms: Dexmedetomidine; ephedrine; midazolam; propofol
Drug: midazolam — All patients were premedicated with midazolam 0.02 mg/kg before induction.
  Arms: midazolam
Drug: propofol — All patients in both groups received a bolus dose of propofol 0.3 mg/kg for sedative effect.
  Other Names: Pofol
  Arms: propofol
Drug: ephedrine — Ephedrine 5 mg was injected when systolic blood pressure decreased below 90 mmHg
  Arms: ephedrine

SUMMARY:
This randomised, double-blind study compared remifentanil and dexmedetomidine for monitored anaesthesia care (MAC) during minimally invasive corrections of vertebral compression fracture (vertebroplasty (VP) and kyphoplasty (KP)).

In total, 80 ASA physical status I-III patients scheduled for VP and KP randomly received remifentanil or dexmedetomidine to maintain OAA/S scale ≤ 4 during the procedures. Multiple hemodynamic variables of patients were recorded and the frequency of oxygen desaturation, respiratory depression, intraoperative need for other opioids, recovery time, operator satisfaction score, and patients' overall pain experiences were also compared.

The investigators are expecting that both remifentanil and dexmedetomidine appear to be quite safe for MAC during VP and KP. Thus, dexmedetomidine may be an alternative for MAC during VP and KP in elderly patients.

DETAILED DESCRIPTION:
All patients fasted for 8 h before the procedure and were premedicated with midazolam 0.02 mg/kg. In the prone position, patients were monitored by ECG, non-invasive blood pressure, and pulse oximetry, and received supplemental oxygen (3 L/min) via a nasal cannula during the procedure.

Study drugs were prepared in 20 mL and 50 mL syringes to maintain a double-blind design. One anaesthesiologist administered normal saline or dexmedetomidine contained in the 20-mL syringe during the initial 10 min for loading dose of dexmedetomidine. Then, another investigator who did not know which syringes contained remifentanil or dexmedetomidine adjusted the infusion rate with a 50-mL syringe according to patients' response. After all patients in both groups received a bolus dose of propofol 0.3 mg/kg, patients given remifentanil received continuous infusion of the drug at 1-5 µg/kg/h, and patients receiving dexmedetomidine were given that drug at 0.3-0.4 µg/kg over 10 min, followed by continuous infusion of dexmedetomidine 0.2-1 µg/kg/h throughout the procedure. Levels of patient sedation were checked during the procedure and infusion rates of the study drugs were adjusted to maintain alertness/sedation below 4 on the OAA/S scale.

Mean arterial pressure (MAP), heart rate (HR), oxygen saturation (SpO2), respiratory rate (RR), and adverse effects of the study drugs were recorded during the procedure. Ephedrine 5 mg was injected when systolic blood pressure decreased below 90 mmHg. Duration of PACU stay was also recorded.

Operator satisfaction score and patient's overall pain experience were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled for vertebroplasty or kyphoplasty under monitored anesthesia care
* ASA status I-III
* aged more than 65 years old.

Exclusion Criteria:

* obesity (BMI > 30 kg/m2)
* hypotension (systolic blood pressure < 100 mmHg)
* bradycardia (heart rate < 60 bpm)
* heart block
* baseline oxygen desaturation (SpO2 < 90%)
* sleep apnea
* asthma, or chronic obstructive pulmonary disease
* those who refused to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The frequencies of oxygen desaturation during procedures | About 1 hour through the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Eun Young Park, MD, Study Chair — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Dongan-gu, South Korea

REFERENCES:
- [Background] Nevitt MC, Ettinger B, Black DM, Stone K, Jamal SA, Ensrud K, Segal M, Genant HK, Cummings SR. The association of radiographically detected vertebral fractures with back pain and function: a prospective study. Ann Intern Med. 1998 May 15;128(10):793-800. doi: 10.7326/0003-4819-128-10-199805150-00001. PMID 9599190
- [Background] Sen J, Sen B. A comparative study on monitored anesthesia care. Anesth Essays Res. 2014 Sep-Dec;8(3):313-8. doi: 10.4103/0259-1162.143121. PMID 25886327
- [Background] Ryu JH, Lee SW, Lee JH, Lee EH, Do SH, Kim CS. Randomized double-blind study of remifentanil and dexmedetomidine for flexible bronchoscopy. Br J Anaesth. 2012 Mar;108(3):503-11. doi: 10.1093/bja/aer400. Epub 2011 Dec 15. PMID 22174346
- [Background] Holas A, Krafft P, Marcovic M, Quehenberger F. Remifentanil, propofol or both for conscious sedation during eye surgery under regional anaesthesia. Eur J Anaesthesiol. 1999 Nov;16(11):741-8. doi: 10.1046/j.1365-2346.1999.00574.x. PMID 10713867
- [Background] Hsu YW, Cortinez LI, Robertson KM, Keifer JC, Sum-Ping ST, Moretti EW, Young CC, Wright DR, Macleod DB, Somma J. Dexmedetomidine pharmacodynamics: part I: crossover comparison of the respiratory effects of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1066-76. doi: 10.1097/00000542-200411000-00005. PMID 15505441
- [Background] Mohr M, Pillich D, Kirsch M, Mueller JU, Fleck S, Hosten N, Langner S. Percutaneous balloon kyphoplasty with the patient under intravenous analgesia and sedation: a feasibility study. AJNR Am J Neuroradiol. 2011 Apr;32(4):649-53. doi: 10.3174/ajnr.A2345. Epub 2011 Jan 27. PMID 21273350
- [Background] Della Puppa A, Andreula C, Frass M. Assisted sedation: a safe and easy method for pain-free percutaneous vertebroplasty. Minerva Anestesiol. 2008 Mar;74(3):57-62. PMID 18288067
- [Derived] Lee JM, Lee SK, Lee SJ, Hwang WS, Jang SW, Park EY. Comparison of remifentanil with dexmedetomidine for monitored anaesthesia care in elderly patients during vertebroplasty and kyphoplasty. J Int Med Res. 2016 Apr;44(2):307-16. doi: 10.1177/0300060515607385. Epub 2016 Feb 18. PMID 26912506